CLINICAL TRIAL: NCT07370857
Title: The Effect of Music Medicine on Anxiety and Pain Levels in Women Undergoing Embryo Transfer: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, helin kalır, PhD Candidate, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hasan Kalyoncu
Record Dates: First submitted 2025-12-17; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-05

CONDITIONS: Pain Management; Infertility (IVF Patients); Anxiety
MeSH Terms: conditions — Agnosia; Infertility; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 1. Music Medicine Group (Arm 1) Label: Music Medicine Group
     Arm Type: Experimental
     Description: Participants listen to patient-selected music via noise-canceling headphones throughout the embryo transfer procedure and for 15 minutes post-procedure, in addition to standard care.
  2. Control Group (Arm 2) Label: Control Group
  Arm Type: No Intervention
  Description: Participants receive standard clinical care for the embryo transfer procedure without any music medicine intervention.
Who Masked: Participant
Masking Description: Randomization was performed using the sealed envelope method to ensure allocation concealment; therefore, the investigator did not know the group assignments until the point of intervention. Due to the nature of the music medicine intervention, the participants and the investigator collecting the data could not be masked during the procedure. However, to minimize bias, the statistical analysis will be conducted by a researcher blinded to the group allocations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Medicine Group (Experimental): Patients in this group receive music medicine intervention in addition to standard care during the embryo transfer process.
  Interventions: Behavioral: "Patient-Selected Music Medicine
- Control Group (No Intervention): Participants receive only the standard clinical procedures and routine care for embryo transfer without any music intervention.

INTERVENTIONS:
Behavioral: "Patient-Selected Music Medicine — Participants in the intervention group listen to their pre-selected music through high-quality, over-ear active noise-canceling headphones to ensure acoustic isolation. The music intervention begins immediately before the embryo transfer, continues throughout the procedure, and extends for 15 minutes in the recovery room. The volume is adjusted by the patient to a comfortable level, and disposable covers are used on the headphones for hygiene.
  Arms: Music Medicine Group

SUMMARY:
This study was designed to investigate the effects of music medicine on anxiety, pain, and vital signs in women undergoing embryo transfer. The study followed a randomized controlled design and was conducted at the IVF unit of a university hospital. The sample consisted of women who met the specified inclusion criteria, and participants were assigned to the intervention and control groups using randomization.

Data collection tools included a socio-demographic characteristics form, a vital signs recording form (blood pressure, pulse, respiratory rate, and oxygen saturation), the State-Trait Anxiety Inventory (STAI-I and II), and the Visual Analogue Scale (VAS). The intervention group listened to patient-selected music during the embryo transfer process, while the control group received standard care. Measurements were taken before, during, and after the embryo transfer.

The obtained data were analyzed using appropriate statistical methods to evaluate the effects of music on anxiety, pain levels, and vital signs. This study aims to improve women's embryo transfer experiences by contributing to nursing care and reproductive health practices.

DETAILED DESCRIPTION:
The study evaluates the effect of music medicine on anxiety and pain levels during embryo transfer. Participants in the intervention group listen to patient-selected music via noise-canceling headphones. The process includes baseline assessments of vital signs and anxiety, followed by post-intervention measurements 15 minutes after the procedure.

ELIGIBILITY:
Inclusion Criteria:

Women undergoing embryo transfer.

Ages 18 to 45 years (or your specific age range).

Literacy in Turkish to complete the inventories.

Voluntarily agreeing to participate in the study.

Exclusion Criteria:

Patients with hearing impairment.

Patients with cognitive or psychiatric disorders that prevent completion of the inventory.

Patients who have taken analgesic or anxiolytic medication within the last 24 hours.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
State Anxiety Score | Measured at two time points: baseline (pre-test, upon admission to the room) and 15 minutes after the embryo transfer procedure (post-test).
  Measured using the Spielberger State-Trait Anxiety Inventory (STAI). Only the "State" subscale is used to assess the current level of anxiety related to the embryo transfer procedure. The score ranges from 20 to 80, where higher scores indicate higher levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Harran University, Sanliurfa, Şanlıurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared to protect participant privacy and because the data are currently being used as part of a doctoral dissertation. Results will be disseminated through publication in peer-reviewed journals.